CLINICAL TRIAL: NCT02502526
Title: Comparison of Cumulative Dissipated Energy (CDE) and Balanced Salt Solution (BSS) Fluid Used With the Centurion® With the 45° Degree Balanced Ultrasound (U/S) Tip vs the Centurion® With Mini Flared Kelman U/S Tip vs the Infiniti® With Mini Flared Kelman U/S Tip on Hard Lenses
Brief Title: Comparison of Centurion® Vision System With Balanced Tip and the Infiniti® Vision System With the Mini Flared Kelman (MFK) Tip During Cataract Extraction Surgery of Hard Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTU424-P001
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-04

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — Chorionic Villi Sampling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CVS with 45° Balanced Tip (Experimental): Centurion® Vision System, 45° Balanced Tip used with INTREPID® Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
  Interventions: Device: Centurion® Vision System, 45° Balanced Tip; Device: INTREPID® Ultra infusion sleeve
- CVS with 45° MFK Tip (Active Comparator): Centurion® Vision System, 45° MFK Tip used with INTREPID® Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
  Interventions: Device: Centurion® Vision System, 45° MFK Tip; Device: INTREPID® Ultra infusion sleeve
- IVS with 45° MFK Tip (Active Comparator): lnfiniti® Vision System, 45° MFK Tip used with Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
  Interventions: Device: lnfiniti® Vision System, 45° MFK Tip; Device: Ultra infusion sleeve

INTERVENTIONS:
Device: Centurion® Vision System, 45° Balanced Tip
  Other Names: CVS with 45° Balanced Tip
  Arms: CVS with 45° Balanced Tip
Device: Centurion® Vision System, 45° MFK Tip
  Other Names: CVS with 45° MFK Tip
  Arms: CVS with 45° MFK Tip
Device: lnfiniti® Vision System, 45° MFK Tip
  Other Names: IVS with 45° MFK Tip
  Arms: IVS with 45° MFK Tip
Device: INTREPID® Ultra infusion sleeve
  Arms: CVS with 45° Balanced Tip; CVS with 45° MFK Tip
Device: Ultra infusion sleeve
  Arms: IVS with 45° MFK Tip

SUMMARY:
The purpose of this study is to demonstrate that the Centurion® Vision System (CVS) used with the 45° Balanced Tip will result in less Cumulative Dissipated Energy (CDE) than the lnfiniti® Vision System (IVS) used with the 45° Mini-Flared Kelman (MFK) tip during cataract extraction surgery via phacoemulsification of cataract grades NII- NIV [Lens opacities classification system II (LOCSII)].

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to consent for participation;
* Willing and able to attend postoperative examinations per protocol schedule;
* Cataract in at least one eye with a Nuclear Opalescence of II-IV (via LOCSII) followed by posterior chamber intraocular lens (IOL) implantation;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Planned multiple procedures, including Laser Phaco, LASIK, LRI's etc. during surgery or the course of this study;
* Severe conditions of acute or chronic diseases or illnesses that would increase the operative risk or confound the result of this investigation;
* Untreated or uncontrolled Glaucoma;
* Previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes;
* Poorly dilating pupil or other pupil defect;
* Current or previous use of an alpha-1-selective adrenoceptor blocking agent or antagonist of alpha 1A adrenoceptor (eg, Flomax®, Hyntrin®, or Cardura®);
* Severe retinal disorders;
* Corneal disease or retinal detachment;
* Other protocol-specified exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 study centers located in the United States (2), Hungary (1), and India (1).
Pre-assignment Details: Of the 231 subjects enrolled, 49 were exited prior to randomization (34 due to randomization suspension, 14 due to screen failure, and 1 due to subject death). This reporting group includes all randomized subjects (182).
Groups:
- CVS Bal: Centurion® Vision System (CVS), 45° Balanced Tip used with INTREPID® Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
- CVS MFK: CVS, 45° MFK Tip used with INTREPID® Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
- IVS MFK: lnfiniti® Vision System (IVS), 45° MFK Tip used with Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
Period: Overall Study
Arm/Group | CVS Bal | CVS MFK | IVS MFK
Started (All randomized subjects) | 62 | 59 | 61
Intent-to-Treat (ITT) (All randomized subjects who completed a procedure) | 57 | 57 | 59
Completed (All subjects who completed the study) | 56 | 55 | 55
Not Completed | 6 | 4 | 6
Not completed — Lost to Follow-up | 2 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Disqualified due to cataract grading | 0 | 0 | 1
Not completed — Enrollment suspension | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- CVS Bal: CVS, 45° Balanced Tip used with INTREPID® Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
- IVS MFK: IVS, 45° MFK Tip used with Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
- Total: Total of all reporting groups
Arm/Group | CVS Bal | CVS MFK | IVS MFK | Total
Number analyzed (Participants) | 57 | 57 | 59 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.4) | 70.3 (9.2) | 73.4 (9.6) | 71.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 36 | 98
  Male | 27 | 25 | 23 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 31 | 30 | 89
  Not Hispanic or Latino | 29 | 26 | 29 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Dissipated Energy (CDE)
Description: Cumulative Dissipated Energy (CDE) represents the energy dissipated of the u/s tip and infusion sleeve at the incision point (5.6mm back from the cutting edge of the tip) during the removal of cataractous lens. CDE was reported on the Vision System interface and measured in percent-seconds. A lower CDE indicates that less energy was present at the incision site. Only one eye (study eye) contributed to the analysis. This outcome measure was pre-specified for CVS Bal and IVS MFK.
Time Frame: Day 0 (operative day)
Population: ITT with non-missing data
Measure: Mean (Standard Deviation); unit: percent-seconds
Groups:
- IVS MFK: lVS, 45° MFK Tip used with Ultra Infusion Sleeve in one time routine surgical procedure followed by 3 months (+/- 14 days) of post-operative follow-up
Arm/Group | CVS Bal | IVS MFK
Number analyzed (Participants) | 57 | 58
percent-seconds | 6.2 (2.9) | 11.4 (8.4)
Statistical Analysis 1: Comparison: CVS Bal vs IVS MFK; Test type: Superiority; p < .001, ANCOVA

2. Secondary Outcome: Cumulative Dissipated Energy (CDE)
Description: Cumulative Dissipated Energy (CDE) represents the energy dissipated of the u/s tip and infusion sleeve at the incision point (5.6mm back from the cutting edge of the tip) during the removal of cataractous lens. CDE was reported on the Vision System interface and measured in percent-seconds. A lower CDE indicates that less energy was present at the incision site. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 0 (operative day)
Population: ITT with non-missing data
Measure: Mean (Standard Deviation); unit: percent-seconds
Arm/Group | CVS Bal | CVS MFK | IVS MFK
Number analyzed (Participants) | 57 | 57 | 58
percent-seconds | 6.2 (2.9) | 11.6 (7.3) | 11.4 (8.4)
Statistical Analysis 1: Comparison: CVS Bal vs CVS MFK; Test type: Superiority; p < .001, ANCOVA
Statistical Analysis 2: Comparison: CVS MFK vs IVS MFK; Test type: Superiority; p = 0.605, ANCOVA

3. Secondary Outcome: Balanced Salt Solution (BSS) Fluid Used
Description: BSS Fluid was measured by weighing the BSS bag after priming. BSS Used is Incision Leakage Fluid plus Aspiration Fluid Used. A reduction in BSS fluid used implies less induced trauma to tissues. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 0 (operative day)
Population: ITT with non-missing data
Measure: Mean (Standard Deviation); unit: milliliters (ml)
Arm/Group | CVS Bal | CVS MFK | IVS MFK
Number analyzed (Participants) | 57 | 57 | 58
milliliters (ml) | 95.8 (33.1) | 101.7 (34.3) | 94.1 (34.9)
Statistical Analysis 1: Comparison: CVS Bal vs IVS MFK; Test type: Superiority; p = 0.520, ANCOVA
Statistical Analysis 2: Comparison: CVS MFK vs IVS MFK; Test type: Superiority; p = 0.817, ANCOVA

ADVERSE EVENTS:
Time Frame: Surgery through planned study completion, an average of 3 months
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational product. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Analysis population includes all randomized subjects for whom the procedure was attempted (Safety Analysis Set).
Groups:
- CVS Bal: Subjects exposed to CVS, 45° Balanced Tip
- CVS MFK: Subjects exposed to CVS, 45° MFK Tip
- IVS MFK: Subjects exposed to lVS, 45° MFK Tip
Arm/Group | CVS Bal | CVS MFK | IVS MFK
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/57 | 3/59
Other Adverse Events (participants affected / at risk) | 14/57 | 17/57 | 11/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVS Bal (N=57) | CVS MFK (N=57) | IVS MFK (N=59)
Posterior capsule rupture (Eye disorders) | 1 | 0 | 0
Vitreous loss (Eye disorders) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vitrectomy (Surgical and medical procedures) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CVS Bal (N=57) | CVS MFK (N=57) | IVS MFK (N=59)
Corneal endothelial cell loss (Eye disorders) | 14 | 17 | 11 — Inclusive of any cell loss >20% or under 1,500 cells/mm^2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT02502526/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT02502526/SAP_001.pdf